CLINICAL TRIAL: NCT06952634
Title: A Phase 1, Open Label, Single Dose Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics of ESK001
Brief Title: An Investigational Study of ESK-001 in Participants With Normal Liver Function and Participants With Mild, Moderate, and Severe Liver Damage
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alumis Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESK-001-022
Record Dates: First submitted 2025-04-22; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Healthy Volunteer (Experimental): Up to 24 healthy volunteer participants will receive a single dose of ESK-001
  Interventions: Drug: ESK-001
- Mild Hepatic Impairment (Experimental): 8 participants with mild hepatic impairment will receive a single dose of ESK-001
  Interventions: Drug: ESK-001
- Moderate Hepatic Impairment (Experimental): 8 participants with moderate hepatic impairment will receive a single dose of ESK-001
  Interventions: Drug: ESK-001
- Severe Hepatic Impairment (Experimental): 8 participants with severe hepatic impairment will receive a single dose of ESK-001
  Interventions: Drug: ESK-001

INTERVENTIONS:
Drug: ESK-001 — Single oral dose of ESK-001 in participants from all cohorts

SUMMARY:
This a phase 1, open label, single dose, parallel cohort study to determine the pharmacokinetics (PK) of study drug (ESK-001) in healthy volunteer participants, and participants with mild, moderate, and severe hepatic impairment.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.)

ELIGIBILITY:
Key Inclusion Criteria for All Participants:

* Body mass index between 18.0 and 40.0 kg/m2

Key Inclusion Criteria for Participants with Hepatic Impairment:

* Diagnosis of chronic (> 6 months), stable hepatic impairment with no clinically significant changes within 30 days prior to dosing, as determined by medical history

Key Exclusion Criteria for All Participants:

* Uncontrolled treated/untreated hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 105 mmHg), or uncontrolled treated/untreated hypotension (systolic blood pressure < 90 mmHg and/or diastolic blood pressure < 50 mmHg), or resting pulse rate < 45 or > 100 bpm. Measurements may be repeated once in order to determine eligibility

Key Exclusion Criteria for Healthy Volunteer:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator or designee.
* Positive hepatitis panel and/or positive human immunodeficiency virus test.

Key Exclusion Criteria for Participants with Hepatic Impairment:

* History of any uncontrolled or unstable renal, hematological, gastrointestinal, neurological, endocrine, or psychiatric disorder, as determined by the investigator or designee, within 6 months prior to screening.
* History or current diagnosis of uncontrolled or significant cardiac disease indicative of a significant risk of safety for participation in the study.
* Liver function tests outside the appropriate reference ranges that are not consistent with hepatic dysfunction, as determined by the investigator or designee.
* QTcF > 480 ms for males or > 490 ms for females at screening or check-in, as confirmed from the mean of the original value and 2 repeats.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | 48 hours
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-T)] | 48 hours
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] | 48 hours

SECONDARY OUTCOMES:
Incidence of nonserious adverse events (AE), serious adverse events (SAE), and AE leading to discontinuation | 48 hours
Number of clinically significant changes in clinical laboratory values, vital signs, ECGs, and physical examinations | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jorn Drappa, Medical Director, Study Director — Alumis Inc
Locations (4):
- United States (4):
  - Orange County Research Center, Lake Forest, California
  - Panax Clinical Research, Miami Lakes, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Alliance for Multispecialty Research, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided
The Sponsor Alumis Inc. is a clinical-stage pharmaceutical company that has not yet adopted an Individual Participant Data (IPD) sharing plan.